CLINICAL TRIAL: NCT07363928
Title: A Randomised Controlled Feasibility Study of a Digital Cognitive Behavioural Therapy for Insomnia Intervention in Mild Cognitive Impairment and Mild Dementia: The Randomised Evaluation of Sleep in Cognitive Impairment Trial
Brief Title: A Digital Cognitive Behavioural Therapy for Insomnia Intervention in Mild Cognitive Impairment and Mild Dementia
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24079
Record Dates: First submitted 2026-01-02; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dementia; Mild Cognitive Impairment; Insomnia; Sleep
Keywords: Digital cognitive behavioural therapy for insomnia; dementia; mild cognitive impairment; insomnia; sleep
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: REST is an investigator-blinded, randomised, controlled, two arm, parallel, feasibility study. Participants will be randomised to intervention versus true wait-list control in a 1:1 ratio using a centrally administered, computer-generated randomisation scheme. An asymptotic maximal randomisation strategy, with a maximum tolerated imbalance of three, will be employed. Participants allocated to the intervention group will undertake the digital cognitive behavioural therapy programme (Sleepio). The study co-ordinator will be unblinded to study group assignment in order to facilitate provision of training regarding use of the intervention to those participants assigned to the intervention group. Site investigators, data collectors and statisticians will remain blinded to study group assignment.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants allocated to the intervention group will be provided with access to Sleepio, a fully-automated digital cognitive behavioural therapy for insomnia programme designed to treat insomnia using a combination of evidence-based cognitive and behavioural techniques. Underlying algorithms organise the delivery of information, support, and advice in a manner tailored to each individual participant based on their responses to an initial sleep study questionnaire and subsequent sleep diary entries throughout the duration of the programme.
  The Sleepio programme consists of six sessions, each ranging from five-to twenty minutes in duration. After the first session, each subsequent session is 'unlocked' one week after delivery of the prior session. Accordingly, the programme can be completed within a six-week period. However, the average time taken to complete the programme is 9-10 weeks.
  Interventions: Other: Digital cognitive behavioural therapy for insomnia
- Control Group (No Intervention): Participants allocated to the control group will continue to receive 'treatment-as-usual' throughout the duration of the study period. They will be informed that they will be provided with access to the intervention at the end of the study period.

INTERVENTIONS:
Other: Digital cognitive behavioural therapy for insomnia — Sleepio is a digital cognitive behavioural therapy for insomnia programme designed to treat insomnia by relying on underlying algorithms to tailor delivery of evidence-based cognitive and behavioural techniques based on participants' responses to an initial sleep study questionnaire and subsequent sleep diary entries throughout the duration of the programme.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to assess the feasibility of conducting a definitive randomised controlled trial that will determine the effectiveness of a digital cognitive behavioural therapy for insomnia intervention (Sleepio) in improving sleep, psychosocial health and cognitive performance in people with Mild Cognitive Impairment or mild dementia and co-morbid sleep disturbance.

DETAILED DESCRIPTION:
Sleep is essential to maintain good physical and mental health and plays a central role in many physiological functions. Nevertheless, insomnia is common with approximately one-third of all adults experiencing insomnia symptoms, increasing to 75% in those aged over 65 years. Two recent meta-analyses suggest that insomnia increases the risk of developing dementia.

Cognitive behavioural therapy for insomnia (CBT-I) is the first-line treatment recommended for insomnia and is supported by a large evidence base. Unfortunately, however, CBT-I is often difficult to access due to the shortage of trained therapists. Digital CBT-I (dCBT-I) provides a possible solution to overcome the barriers associated with accessing the traditional therapist-delivered model of CBT-I. There is good evidence regarding the effectiveness of dCBT-I, which has also recently been shown to be feasible and effective in older people. A small mixed-methods study involving 12 participants has demonstrated preliminary acceptability of dCBT-I among older people with Mild Cognitive Impairment (MCI).

Sleepio is a dCBT-I programme that is specifically recommended as first-line treatment for insomnia by the National Institute for Health and Care Excellence (NICE). Underlying algorithms organise the delivery of evidence-based cognitive and behavioural techniques in a manner tailored to each individual based on their responses to an initial sleep study questionnaire and subsequent sleep diary entries throughout the duration of the programme. The Sleepio programme consists of six sessions. The programme can be completed within a six-week period. However, the average time taken to complete the programme is 9-10 weeks.

The investigators aim to conduct a randomised controlled feasibility study of this NICE-recommended dCBT-I intervention in participants with MCI and mild dementia.

Study participants will be community-dwelling adults aged fifty years and older with insomnia and established MCI or mild dementia. All patients attending outpatient memory clinics affiliated with the Mercy University Hospital in Cork City in the south of Ireland will be screened for eligibility. Consecutive patients who meet eligibility criteria will be invited to participate in the study. Where possible, study partners, being close friends or family members of study participants, will be recruited to support participants throughout the study.

Fully informed written consent will be obtained from each participant prior to enrolling them in the study. All participants will be determined able to provide informed written consent as adjudged by a consultant physician in geriatric medicine. Consent will also be obtained from their respective study partners (caregivers/friends/family members) if available and willing to participate.

Participants will be randomised to intervention versus true wait-list control in a 1:1 ratio using a centrally administered, computer-generated randomisation scheme. The study co-ordinator will be unblinded to study group assignment in order to facilitate provision of training regarding use of the intervention to those participants allocated to the intervention group. Site investigators, data collectors and statisticians will remain blinded to study group allocation.

At baseline, upon enrolment in the study, all participants will undergo assessments of their sleep, psychosocial health, cognition and function. These assessments will be repeated at follow up after 10 weeks.

This randomised controlled feasibility study will analyse the feasibility, acceptability and preliminary efficacy of a dCBT-I intervention to improve sleep, psychosocial health and cognitive function in participants with MCI and mild dementia. If shown to be feasible, the results will inform the design of a future definitive randomised controlled trial of the intervention in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years.
2. Sleep Condition Indicator Score ≤16/32.
3. Established Mild Cognitive Impairment (MCI) or mild dementia, diagnosed by a consultant physician specialised in cognitive disorders prior to enrolment in the study. Dementia will be defined using DSM-5 classification and staged according to the Reisberg FAST scale into early/mild stage (Stages 1-4). MCI will be defined using Petersen's criteria. To participate those with MCI/mild dementia must score:

   1. ≥18 on the Mini-Mental State Examination (MMSE), and
   2. ≥0.5-1.0 on the Clinical Dementia Rating (CDR) scale.
4. Internet access for the duration of the intervention (via computer/tablet/smartphone).
5. Sufficient physical/sensory (visual/hearing) capacity to use the intervention, as judged by the clinician/investigator.
6. English-speaker (intervention only available in English).
7. Community-dwellers (non-institutionalised).

Exclusion Criteria:

1. Known history of an International Classification of Diseases (ICD) defined sleep disorder other than insomnia disorder.
2. Receipt of a sleep-related cognitive behavioural therapy (CBT) intervention within the past six months.
3. MMSE score <18 at enrolment, to facilitate adherence and ensure recruitment of those with mild-stage disease.
4. Severe depression (defined as depression requiring hospitalisation in the past 12-months or visit to psychiatry outpatient clinic in the past 3 months).
5. Unstable depression/anxiety disorders or panic attacks (unstable will be defined as changes in antidepressant medications within the last 3 months, i.e. no start, stop or change in dose).
6. Other relevant major neuropsychiatric disorders, including schizophrenia, psychosis, mania, bipolar affective disorder, epilepsy or seizure disorder.
7. Ongoing substance or alcohol abuse.
8. Long-term physical or sensory impairment, pain or other medical condition which, in the opinion of the principal investigator, could impair participation for reasons other than cognitive impairment.
9. Planned surgery or hospitalisation during the study that could interfere with participation.
10. Medical conditions rendering the patient too unwell to continue to participate in the study in the opinion of the principal investigator.
11. A change in the following medication within the three months prior to enrolment:

    1. Benzodiazepine and non-benzodiazepine hypnotic or anxiolytics agents
    2. Cholinesterase inhibitors or Memantine
    3. Antidepressants
    4. Antipsychotics
    5. Amphetamine derivatives
    6. Decongestants (pseudoephedrine, phenylephrine, phenyl¬propanolamine)
    7. Narcotic analgesics
    8. β-Blockers
    9. Pulmonary medications (theophylline and albuterol)
    10. Melatonin

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Participant Recruitment | Six Month Study Period
  The aim of this study is to determine the feasibility of conducting a definitive randomised controlled trial. This primary outcome will assess recruitment of the target number of 30 eligible participants during the six-month study period.
Participant Retention | Six Month Study Period
  The purpose of this study is to determine the feasibility of conducting a definitive randomised controlled trial. This primary outcome will assess retention of the target number of 70% of enrolled participants throughout the study period.
Participant Adherence | Six Month Study Period
  The purpose of this study is to determine the feasibility of conducting a definitive randomised controlled trial. This primary outcome will assess whether participants allocated to the intervention group achieve the target of 66% adherence to the intervention, defined as completion of four out of the six sessions involved in the intervention programme.
Acceptability of the Intervention | Six Month Study Period
  The purpose of this study is to assess the feasibility of conducting a definitive randomised controlled trial. This primary outcome will assess the acceptability of the intervention among the study population using a bespoke questionnaire incorporating the System Usability Scale adapted for cognitive impairment (targeting >70% participants allocated to the intervention group scoring >70/100) and the Usability Metric for User Experience - Lite (UMUX -Lite).
  The System Usability Scale is a validated and commonly employed 10-item Likert-type scale that provides a global assessment of how user-friendly a system or product is perceived to be. The UMUX-Lite is a more condensed 2-item Likert-type scale that also measures user-satisfaction with a system or product.

SECONDARY OUTCOMES:
Sleep - Insomnia Severity Index (ISI) | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in sleep will be assessed using the Insomnia Severity Index (ISI).
  The ISI is a validated 7-item instrument to assess self-reported insomnia severity over the previous two weeks. Scores range from 0-28, with scores greater than or equal to 8 indicating sub-threshold insomnia and scores greater than or equal to 15 indicating clinical insomnia.
Sleep - Sleep Condition Indicator (SCI) | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in sleep will be measured using the Sleep Condition Indicator (SCI).
  The SCI is an 8-item scale validated to assess insomnia based on DSM-5 criteria. Scores range from 0-32, with scores less than or equal to 16 indicating insomnia.
Psychosocial Health - Patient Health Questionnaire 8 (PHQ-8) | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in psychosocial health will be assessed using the Patient Health Questionnaire 8 (PHQ-8), a valid diagnostic and severity measure for depressive disorders.
Psychosocial Health - Generalised Anxiety Disorder 7 (GAD-7), | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in psychosocial health will be measured using the Generalised Anxiety Disorder 7 (GAD-7), a widely-used and validated measure for assessing generalised anxiety disorder.
Psychosocial Health - Euroqol EQ 5D Visual Analogue Scale | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in psychosocial health will be measured using the Euroqol EQ 5D Visual Analogue Scale, which records subjective assessment of health-related quality of life on a 100-point vertical visual analogue scale on which the endpoints are labelled 'the best health you can imagine' and 'the worst health you can imagine'.
Psychosocial Health - Dementia Quality of Life Instrument (DEMQOL) | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in psychosocial health will be measured using the Dementia Quality of Life Instrument (DEMQOL), a validated 29-item measure for assessing self-reported quality of life in people with dementia.
Cognition and Function - Mini-Mental State Examination (MMSE) | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in cognition and function will be measured using the Mini-Mental State Examination (MMSE), a widely used measure of cognitive impairment scored from 0-30 with higher scores indicating better cognition.
Cognition and Function - Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog) | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in cognition and function will be measured using the Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog), a validated assessment of cognition involving 11 tasks and scores ranging from 0-70.
Cognition and Function - Clinical Dementia Rating (CDR) scale | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in cognition and function will be measured using the Clinical Dementia Rating (CDR) scale, a commonly used clinician-rating scale of global symptom severity in dementia.
Cognition and Function - Disability Assessment for Dementia (DAD) | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in cognition and function will be measured using the Disability Assessment for Dementia (DAD), a 40-item assessment of functional ability involving personal and instrumental activities of daily living in people with dementia.
Cognition and Function - British Columbia Cognitive Complaints Inventory (BC-CCI) | Baseline (enrollment) and 10 weeks post-enrollment
  Changes in cognition and function will be measured using the British Columbia Cognitive Complaints Inventory (BC-CCI), a brief 6-item assessment of self-reported cognitive difficulties involving concentration, memory, articulation, thinking and problem-solving over the previous seven days. Scores range from 0-18, with higher scores indicating greater perceived cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Rónán O'Caoimh, PhD, Principal Investigator — Mercy University Hospital
Locations (1):
- Mercy University Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarnai K, Henry A, Miller C, Waxmonsky J, Emsley R, Espie C. 0352 Digital cognitive behavioral therapy in treating insomnia in older adulthood: A sub-analysis using individual participant data. Sleep. 2023;46(Supplement_1):A156-A.
- [Background] Kyle SD, Hurry MED, Emsley R, Marsden A, Omlin X, Juss A, Spiegelhalder K, Bisdounis L, Luik AI, Espie CA, Sexton CE. The effects of digital cognitive behavioral therapy for insomnia on cognitive function: a randomized controlled trial. Sleep. 2020 Sep 14;43(9):zsaa034. doi: 10.1093/sleep/zsaa034. PMID 32128593
- [Background] Espie CA, Kyle SD, Williams C, Ong JC, Douglas NJ, Hames P, Brown JS. A randomized, placebo-controlled trial of online cognitive behavioral therapy for chronic insomnia disorder delivered via an automated media-rich web application. Sleep. 2012 Jun 1;35(6):769-81. doi: 10.5665/sleep.1872. PMID 22654196
- [Background] Espie CA, Emsley R, Kyle SD, Gordon C, Drake CL, Siriwardena AN, Cape J, Ong JC, Sheaves B, Foster R, Freeman D, Costa-Font J, Marsden A, Luik AI. Effect of Digital Cognitive Behavioral Therapy for Insomnia on Health, Psychological Well-being, and Sleep-Related Quality of Life: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Jan 1;76(1):21-30. doi: 10.1001/jamapsychiatry.2018.2745. PMID 30264137
- [Background] Hoyos C, Espinosa N, Marshall N, LaMonica H, Gordon C, Rainey-Smith S, et al. 0441 Sleep Disturbance in MCI: A Pilot Study of a Cognitive Behavioural Therapy Digital Intervention (SUCCEED). Sleep. 2024;47(Supplement_1):A189-A.
- [Background] Mattos MK, Manning CA, Quigg M, Davis EM, Barnes L, Sollinger A, Eckstein M, Ritterband LM. Feasibility and Preliminary Efficacy of an Internet-Delivered Intervention for Insomnia in Individuals with Mild Cognitive Impairment. J Alzheimers Dis. 2021;84(4):1539-1550. doi: 10.3233/JAD-210657. PMID 34690141
- [Background] Lee Y, Kim I, Lee S, Yu S. Information and Communication Technology-Based Application for Cognitive Behavioral Therapy among Community-Dwelling Older Adults with Insomnia: Development and Validation Study. Healthcare (Basel). 2024 Jan 2;12(1):106. doi: 10.3390/healthcare12010106. PMID 38201011
- [Background] Zachariae R, Lyby MS, Ritterband LM, O'Toole MS. Efficacy of internet-delivered cognitive-behavioral therapy for insomnia - A systematic review and meta-analysis of randomized controlled trials. Sleep Med Rev. 2016 Dec;30:1-10. doi: 10.1016/j.smrv.2015.10.004. Epub 2015 Oct 24. PMID 26615572
- [Background] Soh HL, Ho RC, Ho CS, Tam WW. Efficacy of digital cognitive behavioural therapy for insomnia: a meta-analysis of randomised controlled trials. Sleep Med. 2020 Nov;75:315-325. doi: 10.1016/j.sleep.2020.08.020. Epub 2020 Aug 26. PMID 32950013
- [Background] Koffel E, Kuhn E, Petsoulis N, Erbes CR, Anders S, Hoffman JE, Ruzek JI, Polusny MA. A randomized controlled pilot study of CBT-I Coach: Feasibility, acceptability, and potential impact of a mobile phone application for patients in cognitive behavioral therapy for insomnia. Health Informatics J. 2018 Mar;24(1):3-13. doi: 10.1177/1460458216656472. Epub 2016 Jun 27. PMID 27354394
- [Background] Naismith SL, Pye J, Terpening Z, Lewis S, Bartlett D. "Sleep Well, Think Well" Group Program for Mild Cognitive Impairment: A Randomized Controlled Pilot Study. Behav Sleep Med. 2019 Nov-Dec;17(6):778-789. doi: 10.1080/15402002.2018.1518223. Epub 2018 Sep 24. PMID 30247939
- [Background] Cassidy-Eagle E, Siebern A, Unti L, Glassman J, O'Hara R. Neuropsychological Functioning in Older Adults with Mild Cognitive Impairment and Insomnia Randomized to CBT-I or Control Group. Clin Gerontol. 2018 Mar-Apr;41(2):136-144. doi: 10.1080/07317115.2017.1384777. Epub 2017 Dec 8. PMID 29220627
- [Background] Crowley P, O'Donovan MR, Leahy P, Flanagan E, O'Caoimh R. Pharmacological and Non-Pharmacological Interventions to Improve Sleep in People with Cognitive Impairment: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2025 Jun 18;22(6):956. doi: 10.3390/ijerph22060956. PMID 40566383
- [Background] Riemann D, Espie CA, Altena E, Arnardottir ES, Baglioni C, Bassetti CLA, Bastien C, Berzina N, Bjorvatn B, Dikeos D, Dolenc Groselj L, Ellis JG, Garcia-Borreguero D, Geoffroy PA, Gjerstad M, Goncalves M, Hertenstein E, Hoedlmoser K, Hion T, Holzinger B, Janku K, Jansson-Frojmark M, Jarnefelt H, Jernelov S, Jennum PJ, Khachatryan S, Krone L, Kyle SD, Lancee J, Leger D, Lupusor A, Marques DR, Nissen C, Palagini L, Paunio T, Perogamvros L, Pevernagie D, Schabus M, Shochat T, Szentkiralyi A, Van Someren E, van Straten A, Wichniak A, Verbraecken J, Spiegelhalder K. The European Insomnia Guideline: An update on the diagnosis and treatment of insomnia 2023. J Sleep Res. 2023 Dec;32(6):e14035. doi: 10.1111/jsr.14035. PMID 38016484
- [Background] Edinger JD, Arnedt JT, Bertisch SM, Carney CE, Harrington JJ, Lichstein KL, Sateia MJ, Troxel WM, Zhou ES, Kazmi U, Heald JL, Martin JL. Behavioral and psychological treatments for chronic insomnia disorder in adults: an American Academy of Sleep Medicine clinical practice guideline. J Clin Sleep Med. 2021 Feb 1;17(2):255-262. doi: 10.5664/jcsm.8986. PMID 33164742